CLINICAL TRIAL: NCT06998576
Title: Different Strokes for Different Folks - Leveraging on Social Networks for Public Health Education on Antibiotic Use and Antimicrobial Resistance
Brief Title: Using Social Influencers for Public Health Education on Antibiotic Use and Antimicrobial Resistance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Chow Li Ping Angela, Senior Consultant, Department of Epidemiology and Preventive Medicine, Tan Tock Seng Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSAINV22jul-0010
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Community Members
Keywords: public health education; antimicrobial resistance; antibiotic use; animated educational video; neighborhood establishments

STUDY DESIGN:
Intervention Model Description: A quasi-experimental study will be conducted to compare the effectiveness of public health education via an animated educational video on antibiotic use and AMR that is facilitated by neighborhood food and beauty establishments (social influencers) with that facilitated through clinics (traditional source of information).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthcare clinics (Experimental): Ten healthcare clinics will be chosen. Patients will enrol into the study by scanning the QR code on the recruitment poster at the participating healthcare clinics will access the health educational intervention.
  Interventions: Behavioral: Animated educational video on antibiotic use
- Food establishments (Experimental): Ten food establishments will be chosen. Patrons will enrol in the study by scanning the QR code on the recruitment poster at the participating F&B shops will access the health educational intervention.
  Interventions: Behavioral: Animated educational video on antibiotic use
- Beauty establishments (Experimental): Ten beauty etablishments will be chosen. Patrons will enrol in the study by scanning the QR code on the recruitment poster at the participating beauty establishments will access the health educational intervention.
  Interventions: Behavioral: Animated educational video on antibiotic use

INTERVENTIONS:
Behavioral: Animated educational video on antibiotic use — The intervention features a concise animated video on antibiotic use and AMR. The video's content and format will be developed based on the results of a survey conducted among the community residents in the two neighborhoods. Through the survey, the participants evaluated multiple message options including the various delivery formats. The animated video was designed incorporating the community's preferred key message and delivery method. The resulting video uses graphics, voice-overs, captions [in all 4 official national languages] to convey key messages about appropriate antibiotic use and AMR.

SUMMARY:
This study aims to compare the effectiveness of health education facilitated by neighborhood food and beauty establishments with that facilitated by clinics in increasing the public's knowledge of antibiotic use and antimicrobial resistance (AMR) and improving antibiotic behaviors.

The quasi-experimental study will involve a total of 3300 patrons of the 10 most popular consenting clinics, food and beauty establishments respectively, in two neighborhoods in Singapore.

Recruitment Process

1. Participants will scan the QR code on the posters in the participating clinics/establishments
2. Read the study information sheet
3. Consent will be implied on submission of survey
4. Total recruitment period: One year
5. Target: 3300 patrons of the 30 establishments (10 each of clinics, food, and beauty establishments)

Intervention Structure

1. Participants will complete a pre-intervention/baseline survey (#1)
2. Intervention includes an animated educational video with key messages on appropriate antibiotic use and AMR
3. Followed by immediate post-intervention survey (#2)
4. Provide contact details (mobile phone number) for reimbursement & future follow-up online surveys
5. Complete follow-up online surveys: at 1 month post-intervention (#3), 3 months post-intervention (#4) and 6 months post-intervention (#5)

Expected Outcomes Increase in public knowledge of antibiotic use and AMR, and antibiotic behaviors through health education facilitated by neighborhood food and beauty establishments, in addition to that facilitated by clinics

DETAILED DESCRIPTION:
According to the World Health Organisation (WHO), antimicrobial resistance (AMR) is one of top 10 global public health threats facing humanity [1,2] and is primarily driven by overuse and misuse of antibiotics [3]. Majority of the population-based national AMR educational campaigns focused on raising public awareness of appropriate antibiotic use and promoting action against antimicrobial resistance have shown mixed results largely due to its "one-size-fits-all" approach [4,5,6].

While healthcare providers are key players in health communication and considered most trusted sources of health information across all age groups [7], there is a need to identify and harness non-healthcare related establishments which can serve as trusted sources of health information especially for younger age groups who are less likely to have healthcare encounters [8-10]. The present study aims to engage non-healthcare establishments (food and beauty) with high degree centrality in the community identified through social network analysis, and evaluate the effectiveness of sharing health information about antibiotic use facilitated by non-healthcare establishments (food and beauty) as compared to traditional healthcare sources (clinics).

The Investigators conducted an exploratory sequential mixed methods study to identify both healthcare and non-healthcare (food and beauty) establishments which were highly frequented by the residents in the community. Findings from the above study were used to select the top 10 highly frequented healthcare and non-healthcare (food and beauty) establishments.

A quasi-experimental study will be conducted to compare the effectiveness of sharing health information about antibiotic use and AMR facilitated through healthcare clinics, and beauty and food establishments in 2 neighborhoods. Participants (patients/patrons) who visit the participating establishments (clinics/food establishments/beauty establishments) will be invited to take part in the study by scanning the QR code on the recruitment posters placed inside the premises. Upon scanning the QR code, participants will proceed to complete a pre-intervention questionnaire survey (#1) on an online platform after going through the study information sheet. Upon completion of the survey #1, participants will be guided through embedded instructions to click on a link to access the health educational intervention. The educational intervention includes a short 2-minute animated video (developed based on the preferences of the community as identified from the results of the quantitative survey) will be hosted on a multimedia online platform providing key information on appropriate antibiotic use and AMR. After viewing the video, the participants will be subsequently led to the post-intervention survey #2 via a link. Before submitting survey #2, contact details (mobile number) and the preferred payment method will be collected for reimbursement purposes and future follow-up surveys. The enrolled participants will be re-contacted by the study team via a mobile messaging service (such as WhatsApp), and will be guided through embedded instructions to complete three more surveys (#3, #4 & #5) at 1-, 3-, and 6-month post-intervention to assess knowledge on antibiotic use and AMR and behaviors on antibiotic use. Participants will be recruited from all 30 participating establishments (10 clinics, 10 F&B shops, 10 beauty salons) for the entire study duration of one year and will be followed up for 6 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21 years and above
* Patrons of the 30 participating healthcare clinics, food and beauty establishments

Exclusion Criteria:

* Patrons who are already enrolled in the study at one of the 30 participating establishments

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3300 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Knowledge of antibiotic use - 3 questions from the World Health Organization's Antibiotic Resistance Multi-country Public Awareness Survey questionnaire | The participants will be followed up for 6 months following the intervention.
  Proportion of participants with good knowledge of antibiotic use at baseline (pre-intervention), immediate post-intervention, and at 1-month, 3-month and 6-month post-intervention.
Knowledge of AMR - 8 questions from the World Health Organization's Antibiotic Resistance Multi-country Public Awareness Survey questionnaire | The participants will be followed up for 6 months following the intervention.
  Proportion of participants with good knowledge of AMR at baseline (pre-intervention), immediate post-intervention, and at 1-month, 3-month and 6-month post-intervention.
Appropriate antibiotic use - 6 questions adapted from the US Centers for Disease Control and Prevention's advisory on appropriate antibiotic use | The participants will be followed up for 6 months following the intervention.
  Proportion of participants who use antibiotics appropriately at baseline (pre-intervention), immediate post-intervention, and at 1-month, 3-month and 6-month post-intervention.

SECONDARY OUTCOMES:
Reach - using the RE-AIM framework | one year study duration for enrollment
  The absolute number and proportion of participants who enrol in the study over the one year duration, and also enrollment rate by establisment type over one year
Implementation fidelity - using the RE-AIM framework | one year study duration for doing fidelity checks
  Monthly physical visits at all 30 participating establishments for checking poster integrity at the premises and whether staff invite patrons to enrol in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chow A, Aithal S, Guo H, Lwin MO, Hildon ZJ. Using social influencers for public health education on antibiotic use and antimicrobial resistance: protocol for a quasi-experimental study. BMC Public Health. 2025 Sep 24;25(1):3120. doi: 10.1186/s12889-025-24338-z. PMID 40993665